CLINICAL TRIAL: NCT02997683
Title: Influence of Training With Whole Body Vibration Device on Quality of Life (QoL), Exercise Capacity, as Well as on the Effects of Muscle Power and Muscle Function in Patients With Pulmonal Arterial Hypertension (PAH) in an Extended 3-month Home Based Training. Background and Rationale for the Proposal: Capacity and the Ability to Exercise, in Patients With PAH is Limited. Primary Scientific Question Addressed:Changes in Muscle Power, Changes in 6-Minute Walk Distance (6MWD) and Changes in QoL Are to be Evaluated.
Brief Title: 3-Month Home-based Training With Whole Body Vibration Device in Patients With PAH (GALILEO-PAH-HOME)
Acronym: GALILEOHOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinikum der Universität Köln (Other)
Responsible Party: Principal Investigator, Felix Gerhardt, Dr. med., Klinikum der Universität Köln
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Changes in Six Minute Walking Distance, Peak Oxygen Uptake, Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-month home based training on whole body vibration platform (Experimental): This Group will receive a training device to perform their given exercises on
  Interventions: Device: Body Vibration platform GALILEO
- 3-month home based training on floor (Placebo Comparator): This Group will perform their given exercises at home on the floor
  Interventions: Other: exercises at home on the floor

INTERVENTIONS:
Device: Body Vibration platform GALILEO — 3 month home based training on whole Body Vibration platform GALILEO
  Arms: 3-month home based training on whole body vibration platform
Other: exercises at home on the floor — exercises at home on the floor
  Arms: 3-month home based training on floor

SUMMARY:
In order to evaluate Long term effects of whole Body Vibration (wbv) in patients with PAH and CTEPH patients will get a training device to use at home for 3 months. Patients in the Intervention group will be introduced in the training program on the wbv-device in the study center 3-4 times and baseline Parameters will be collected before start of the home based training. Patients randomized into the placebo arm be introduced into the training program according to the interventional arm but not perfoming the exercises on the wbv-device but on the floor.

DETAILED DESCRIPTION:
Screening (day -21 until day -7): Subjects will be evaluated according to In- and Exclusion critera

Randomization (day -7): Subjects will be randomized to either Intervention Group (training on wbv platform) or non-Intervention Group (training without wbv).

Introduction Week -1(-7d-d1): All subjects will receive introduction in their training

Month 1:

Day 1: From this day subjects are supposed to start their training accoridng to protocol

Day 2: Telephone Visit

Day 5: Telephone Visit

Day 7: Telephone Visit

Day 10: Telephone Visit

Day 13: Telephone Visit

Day 20: Telephone Visit

Day 27: Telephone Visit

Week 4, Day 28: Study center Visit: 6MWD, QoL-Questionnaire, AEs, re-training

Month 2:

Week 5, Day 34:

Week 6, Day 41:

Week 7, Day 48:

Week 8, Day 55:

Month 3:

Week 9, Day 62:

Week 10, Day 69:

Week 11, Day 76:

Week 12, Day 83: Final Visit

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-90 years
* Signed informed consent
* Symptomatic PAH (idiopathic, hereditary or associated with systemic scleroderma)
* Persistend or inoperable CTEPH
* Invasively confirmed PAH
* 6MWT ≥ 50 - 450 m
* Stable specific therapy for at least 6 weeks
* Ability to perform bike test
* Ability to perform wbv training
* NYHA/WHO-FC II-III

Exclusion Criteria:

any other PAH/PH than idiopathic, hereditary, associated with systemic scleroderma or CTEPH

* Rehabilitation or other training concept performed within 6 weeks before inclusion
* pregnancy
* acute thrombosis
* newly implanted Hip or Knee
* recent bone fracture
* Disability to confirm consent
* NYHA/WHO-FC IV
* 6MWD below 50 or above 450 m

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in 6 Minute Walking distance | 3 months
Changes in 6 Minute Walking distance | 4 weeks interm analysis

SECONDARY OUTCOMES:
Changes in Peak Oxygen uptake in cardiopulmonary exercise testing (CPET) | 3 months
Changes in Peak Oxygen uptake in cardiopulmonary exercise testing (CPET) | 4 weeks
Changes in Quality of Life | 3 months
Changes in Quality of Life | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Spezialambulanz für pulmonale Hypertonie Uniklinik Köln, Cologne, North Rhine-Westphalia, Germany